CLINICAL TRIAL: NCT04785274
Title: The Effect of Non-invasive Hemoglobin Measurement on Blood Transfusion and Mortality in Hip Surgeries: a Randomized Controlled Trial
Brief Title: The Effect of Non-invasive Hemoglobin Measurement in Hip Surgeries
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, OZCAN PISKIN, MD, Clinical Professor, Bulent Ecevit University
Other Study IDs: 2020-24/16/12/2020
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Bleeding; Hemorrhage; Hemodynamic Instability
Keywords: Perioperative Bleeding; Mortality; Hemoglobin; Non-invasive monitoring; Transfusion;; SpHb
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SpHb
  Interventions: Device: non-invasive hemoglobin (SpHb)
- Control
  Interventions: Device: non-invasive hemoglobin (SpHb)

INTERVENTIONS:
Device: non-invasive hemoglobin (SpHb) — hemoglobin measuring device

SUMMARY:
Bleeding is one of the most important causes of mortality and morbidity in patients.

Hb levels are the most prevalently utilized monitoring parameter in hemorrhagic patients in the hemodynamic sense. Hemoglobin determination is studied at laboratories along with blood gasses or complete blood analysis. Recently, non-invasive techniques where measurement is made from the fingertips have been offered for use. One of these techniques is non-invasive hemoglobin (SpHb) measurement. SpHb is used as a trend monitor. Based on the severity of bleeding, the compensatory mechanisms of patients may be disrupted. This situation may lead to lower levels of toleration of anemia during bleeding. The relationship between blood transfusion and mortality is under debate.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* General anesthesia undergoing hip surgery
* American society of anesthesiology (ASA) scores I-II-III

Exclusion Criteria:

* Receiving inotropic support
* Uncontrolled diabetes
* Arrhythmia
* Hypothermia
* Hyperbilirubinemia
* Jaundice
* Dark skin pigmentation
* Without voluntary consent
* Hypovolemia,
* hypotension,
* sepsis,
* blood diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: General anesthesia undergoing hip surgery
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Hemodynamic Stability | during the surgery
  to compare blood transfusion decisions made with SpHb measurement values and with conventional methods in patient who would receive hip surgery.

SECONDARY OUTCOMES:
Mortality | until 3 months after surgery
  to compare the effects of transfusion results on mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bulent Ecevit University Medicine Faculty, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No